CLINICAL TRIAL: NCT04178798
Title: Phase III Randomized Study to Investigate the Use of Acalabrutinib in the Treatment of Patients With Early Stage CLL With High Risk of Early Disease Progression
Brief Title: Study to Investigate the Use of Acalabrutinib in the Treatment of Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLLC-EARLY
Record Dates: First submitted 2019-11-08; First posted 2019-11-26 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Chronic Lymphocytic Leukemia- Binet Staging System
Keywords: CLL
MeSH Terms: interventions — acalabrutinib

STUDY DESIGN:
Intervention Model Description: * Arm A (65 patients): Patients assigned to arm A, will receive acalabrutinib as one capsule of 100 mg orally twice daily on a continuos schedule until disease progression, unacceptable toxicity or early withdrawal.
  * Arm B (65 patients): Patients assigned to arm B, will remain on the w&w approach until disease progression or early withdrawal.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A_Acalabrutinib (Experimental): Patients assigned to arm A, will receive acalabrutinib as one capsule of 100 mg orally twice daily on a continuos schedule until disease progression, unacceptable toxicity or early withdrawal.
  Interventions: Drug: Acalabrutinib 100 MG Oral Capsule
- Arm B_Standard of care (No Intervention): Patients assigned to arm B, will receive standard of care for the management of early Binet stage A patients "clinical observation (watch & wait)" until disease progression or early withdrawal.

INTERVENTIONS:
Drug: Acalabrutinib 100 MG Oral Capsule — Patients in Arm A will receive acalabrutinib as one capsule of 100 mg orally twice daily on a continuos Schedule.
  Arms: Arm A_Acalabrutinib

SUMMARY:
Study Phase III Randomized Study to Investigate the Use of Acalabrutinib in the Treatment of Patients with Early Stage CLL With High Risk of Early Disease Progression.

The study will consist of a screening phase, a treat¬ment/observation phase until progression, and a follow-up phase for progression in patients who discontinue treatment with Acalabrutinib without confirmed progression. Patients who progress will be followed for survival and initiation of subsequent antileukemic therapy. In the study, 130 patients from 20 centers in Spain with intermediate, high or very high risk will be randomized (1:1) to receive Acalabrutinib (n=65) or clinical observation (n=65). Acalabrutinib will be administered orally 100 mg twice daily on a continuous schedule.

Even though the majority of patients with CLL are currently diagnosed at early stages of the disease, there is a consensus that the standard of care in these patients is clinical observation (watch & wait) despite of the presence of risk factors for premature disease progression. Early treatment in patients with adverse prognostic parameters could prevent a disease evolving to a more advanced stage, and therefore more difficult to treat. So far, conventional chemotherapy did not show any benefit in terms of overall survival in patients with early stage CLL. (Dighiero 1998, Hoechstetter Leukemia 2017) Alongside this, treatment with chemotherapy may provoke two undesired effects: first, the occurrence of bone marrow toxicity that may hamper the subsequent administration of other treatments during the course of the disease; second, but not less relevant, genotoxic drug delivery may elicit a phenomenon of clonal selection leading to the appearance of CLL cells with genetic aberrations associated with refractoriness and aggressive outcome (i.e., TP53).

Against this background, it is of interest to investigate the role of new non-genotoxic drugs in the treatment of patients with CLL in early stages. Among different scores for selecting cases that are likely to progress rapidly, the German CLL Study Group (GCLLSG) risk score that includes 8 independent predictors for OS and PFS, differentiates patients with low-risk PFS vs. those with risk of early disease progression (median PFS 87 months vs. less than 27 months), allowing for a risk-adapted treatment approach in early stage CLL. (Pflug 2014, Langerbeins 2015).

Acalabrutinib, a second-generation, selective inhibitor of BTK, has shown substantial activity in patients with CLL. Acalabrutinib is a non-genotoxic drug active in cases with genetic lesions associated with chemorefratoriness and adverse outcome, including patients with alterations of TP53. Therefore, acalabrutinib represents a suitable compound for the treatment of patients with CLL in early stages with risk of early disease progression, including the high-risk CLL patient population with TP53 alterations.

DETAILED DESCRIPTION:
Randomized, open-label, parallel-group, multicenter, phase III trial with two arms, one with acalabrutinib (Arm A) and the other with the standard of care for the management of early Binet stage A patients "clinical observation (watch & wait)" (Arm B) in patients with untreated early stage CLL and risk factors for early disease progression. Early risk of disease progression will be defined by the GCLLSG prognostic index: intermediate (3-5), high (6-10) or very high (11-14) risk scores are required to be included in the study. Randomization will be managed through an IRT system:

* Arm A (65 patients): Patients assigned to arm A, will receive acalabrutinib as one capsule of 100 mg orally twice daily on a continuos schedule until disease progression, unacceptable toxicity or early withdrawal.
* Arm B (65 patients): Patients assigned to arm B, will remain on the w&w approach until disease progression or early withdrawal.

The enrolment period is estimated in 24 months. A treatment cycle is defined as lasting 28 days.

The duration of the study will be of 60 months from the inclusion of the first patient to the last patient has completed the last follow up visit.

1. Periods of patient participation in the study

   * Screening Phase: After providing the written Informed Consent Form (ICF) to participate in the study, patients will be evaluated for eligibility, baseline characteristics and risk factors, during a screening period up to 28 days prior to randomization.
   * Treatment/Observation Phase: The treatment/observation Phase extends from randomization until symptomatic disease progression, unacceptable toxicity or early withdrawal. A treatment cycle is defined as lasting 28 days.
   * Suspected Disease Progression Visit: A visit should be performed at any time when disease progression is suspected. If progression is confirmed, the patient will be followed every 6 months to assess survival status and receipt of subsequent antileukemic therapy until death, patient withdrawal, loss to follow-up, or study termination, whichever comes first. The subsequent treatment decision will be up to the investigator and should generally follow the routine practice.
   * End-of-Treatment/Observation Visit: For patients receiving acalabrutinib, the End-of-Treatment Visit will be performed within 30 days (± 3 days) after the last dose of treatment administration or progression. For patients remaining in the w&w approach, the End-of- Observation Visit will be performed within 30 days of progression.
   * Follow-up for Progression (Pre-PD FU): Patients who discontinue the study treatment without confirmed progression (according to iwCLL guidelines) will continue to be followed for progression every 4 months (±7 days) for the first 24 months of study, then every 6 months (±7 days) until progression or study closure.

   Study visits will no longer be carried out for patients who have withdrawn their informed consent, have died or have been lost to follow-up.
2. Study drug - dosage and administration:

   Acalabrutinib is orally administered and is suitable for formulating in capsules. Acalabrutinib will be supplied by ASTRAZENECA FARMACÉUTICA SPAIN, S.A., on behalf of the Sponsor, as hard gelatin capsules of 100 mg for oral administration. Acalabrutinib can be taken with or without food. As acalabrutinib is metabolized by CYP3A, subjects should be cautioned against using herbal remedies or dietary supplements (in particular, St John's wort, which is a potent CYP3A inducer). Otherwise, subjects should maintain a normal diet unless modifications are required to manage an AE such as diarrhea, nausea or vomiting.
3. Description of Procedures

   * Confirmation of Eligibility: Perform all necessary procedures and evaluations to document that the patient meets each eligibility criterion.
   * Medical History: will include concurrent medical signs and symptoms based upon available documents and patient history.
   * Adverse Events: All medical occurrences that meet the accepted regulatory definition of AE must be recorded from the time the informed consent form is signed until 30 days after the last dose of study drug (in Arm A) or progression (in both arms).
   * Physical Examination, Vital Signs, Height and Weight, ECOG. This will include the lymphatic system, spleen and liver examination as well. will be performed at every visit during the study.
   * Clinical Stage Rai/Binet: A Binet or Rai staging system will be used at every study visit (except on Day 15 Cycle 1 and Day 15 Cycle 2) to stratify patients according to the disease risk.
   * Disease-related symptoms will be assessed and collected at every study visit.
   * Electrocardiogram (ECG) done only at Screening.
   * Concomitant Medication: All medications from 14 days before the start of study drug administration through 30 days after the last dose of study drug or progression.
   * German CLL Study Group (GCLLSG) prognostic index will be determined for each patient only at screening.
   * Cumulative Illness Rating Scale is a measure of comorbid medical conditions that help to characterize patients with concomitant morbidity and fit.
   * Hepatitis Serologies: Hepatitis serologies include Hepatitis C antibody, Hepatitis B surface antigen, Hepatitis B surface antibody, and Hepatitis B core antibody.
   * Hematology: will be performed at every visit by local laboratory and will include a complete blood cell count.
   * Coagulation Panel: Measurement of prothrombin time /INR, and activated partial thromboplastin time will be performed at Screening.
   * Serum chemistry will be locally performed at every visit (except on Day 15 of Cycles 1 and 2)
   * Creatinine clearance (Cockcroft-Gault) will be evaluated (only at screening) by local laboratory.
   * Cytogenetic, CLL FISH Panel within 90 days prior to the inclusion in the study to detect abnormalities in chromosomes 13q, 12, 11q, and 17p must be evaluated.
   * Blood for immunophenotyping (for diagnosis), IGVH mutation status, and serum markers (B2-microglobulin and thymidine kinase) will be centralized in the department of Hematology of the University Hospital of Vall d'Hebron. Blood samples will be collected for all patients at Screening.
   * Serum quantitative immunoglobulin (IgG, IgM, IgA) levels will be evaluated by local laboratory at screening, on Day 1 of every odd cycle from Cycles 3 through 12, on Day 1 of every odd cycle (for Cycles 13, 15, 17, 19, 21 and 23), and then every 3 cycles until progression or study closure.
   * Coombs test will be performed (only at screening) by local laboratory.
   * CT scans of the neck, chest, abdomen, and pelvis.
   * Bone Marrow Aspirate and/or Biopsy should be obtained to confirm CR, or confirm cytopenic progression and distinguish autoimmune versus treatment-related causes. In addition, a further marrow assessment should be performed at any time during follow-up when the patient has cleared MRD from the peripheral blood. Marrow aspirate to confirm CR should have a flow-cytometry-based MRD; MRD should be also analysed in peripheral blood .
   * Overall response assessment will include evaluation of physical exams, recording of symptoms, and hematological evaluations. OR will be assessed on Day 1 Cycle 2, on Day 1 of Cycles 3 to 12, and on Day 1 of Cycles 13, 15, 17, 19, 21, and 23, and then every 3 cycles to disease progression or study closure. For patients in Arm B, response assessment will be performed on Day 1 of every 3 cycles to progression or study termination.
   * Overall Survival: After progression, patients will be followed every 6 months to assess survival status and the start of subsequent cancer therapies until death, patient withdrawal, loss to follow-up, or study termination, whichever comes first.
   * Biomarkers: Blood samples will be collected for an exploratory biomarker assessment at baseline and at progression. Samples at month 3, 6 and 12 will be optional and will collected in patients who have accepted in the inform consent form.
4. Main Efficacy Evaluations Suspected Disease Progression: should be confirmed with a CT scan (or MRI, if CT is contraindicated).

   Disease Evaluation: Objective response will be categorized as CR, CR with incomplete bone marrow recovery (CRi), nodular partial remission (nPR), partial response (PR), stable disease, or progressive disease-all based upon IWCLL criteria (Hallek 2018). Patients who achieve PR in all parameters except lymphocyte count will be considered a PR with lymphocytosis, for the purposes of the Protocol. CRs must be confirmed by bone marrow biopsy/aspirate.

   Given the known mechanism of action of BCR-inhibiting agents, including acalabrutinib, and the treatment-related lymphocytosis frequently observed during treatment with acalabrutinib, isolated treatment-related lymphocytosis (in absence of other clinical, CT, or laboratory evidence of disease progression) will not be considered progressive disease. This approach is supported by the IWCLL guidelines (Hallek 2018).
5. Safety, Monitoring and Reporting: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

   PETHEMA Foundation has delegated Pharmacovigilance functions to the Pharmacovigilance Department of the CRO Dynamic Science S.L.
6. Warnings, Precautions, and Adverse Effects: Acalabrutinib is contraindicated in subjects with clinically significant hypersensitivity to the compound itself or to the excipients in its formulation.

   Hemorrhagic events, including CNS, respiratory, and gastrointestinal hemorrhage, have been reported in clinical trials with acalabrutinib. The mechanism for hemorrhage is not well understood.

   Serious infections, including fatal events, have been reported in clinical studies with acalabrutinib. The most frequently reported Grade 3 or 4 infection was pneumonia. Cases of hepatitis B virus reactivation (resulting in liver failure and death in 1 case) and cases of progressive multifocal leukoencephalopathy have occurred in subjects with hematologic malignancies.

   Cytopenias: treatment-emergent Grade 3 or 4 cytopenias including neutropenia, anemia, and thrombocytopenia have occurred in clinical studies with acalabrutinib.

   Events of second primary malignancies, including non-skin carcinomas, have been reported in clinical studies with acalabrutinib. The most frequently reported was skin cancer.

   Events of atrial fibrillation/flutter have been reported in clinical studies with acalabrutinib, particularly in subjects with cardiac risk factors, hypertension, diabetes mellitus, acute infections, and a previous history of atrial fibrillation. The mechanism for atrial fibrillation is not well understood.

   Subjects should be managed per institutional guidelines with supportive care and diagnostic evaluations as clinically indicated.
7. Drug-drug Interactions: Acalabrutinib is partially metabolized by CYP3A; its exposure is affected when coadministered with strong CYP3A inducers or inhibitors. Consequently, the concomitant use of strong inhibitors/inducers of CYP3A should be avoided when possible. Subjects who require therapy with strong inhibitors of CYP3A should not be enrolled into the study.

   Subjects should avoid the use of calcium carbonate containing drugs or supplements for a period of at least 2 hours before and 2 hours after taking acalabrutinib. Use of omeprazole, esomeprazole, lansoprazole or any other proton pump inhibitors while taking acalabrutinib is not recommended due to a potential decrease in study drug exposure. For subjects who require H2 antagonists, the recommendation is that acalabrutinib is taken at least 2 hours before the H2 antagonist.
8. Treatment-related lymphocytosis, for the purposes of this Protocol, is defined as an elevation in blood lymphocyte count of ≥50% compared to baseline. Acalabrutinib associated treatment-related lymphocytosis generally occurs within the first weeks of therapy, peaks within the first few months, and resolves slowly. Patients with treatment-related lymphocytosis should remain on study treatment and continue with all study-related procedures.
9. Once the complete study is explained, written Informed Consent will be obtained from the patient, legal guardian or representative before starting participation in the study.
10. In order to respect patient privacy, patients will be identified by patient number in all case report forms, study drug accountability logs, study reports and communications. Confidentiality of patients will be kept and their identity will not be disclosed as far as permitted by the law and relevant regulations. Regulation (EU) 2016/679 of the European Parliament and of the Council, of 27 April 2016, on the protection of natural persons with regard to the processing of personal data and the free movement of such data, and Organic Law 3/2018 of December 5, on the Protection or Personal Data and guarantee of digital rights.
11. Early study discontinuation: This study may be discontinued early if, in the Sponsor's opinion, there is sufficient reasonable cause.
12. Data registering and storage: The investigator will keep all study records in compliance with ICH-GCP requirements and current regulations.
13. Responsibility and insurance: The Sponsor has taken out an insurance policy covering, in its terms and conditions, the liability for damages caused to participants and derived from this research, performed fully in compliance with both the scientific Protocol and the applicable law and professional standards.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with previously untreated CLL according to IWCLL criteria (Hallek, 2018).
2. Must understand and voluntarily sign an informed consent form.
3. Age ≥ 18 years at the time of signing the informed consent form and must be able to adhere to the study visit schedule and other Protocol requirements.
4. Diagnosis of CLL prior to inclusion in the study.
5. Binet clinical stage A and Rai 0 or 1.
6. Absence of criteria for the initiation of chemotherapy, defined by the IWCLL guidelines for diagnosis and treatment of CLL (Hallek, 2018):

   * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia.
   * Massive (i.e. ≥6 cm below the left costal margin) or progressive or symptomatic splenomegaly.
   * Massive nodes (i.e. ≥10 cm in longest diameter) or progressive or symptomatic lymphadenopathy.
   * Progressive lymphocytosis with an increase of ≥50% over a 2-month period, or lymphocyte doubling time (LDT) of less than 6 months.
   * A minimum of any one of the following disease-related symptoms: unintentional weight loss ≥10% within the previous 6 months, significant fatigue (i.e., ECOG PS 2 or worse; cannot work or unable to perform usual activities), fevers of ≥38.0°C for 2 or more weeks without other evidence of infection, or night sweats for more than 1 month without evidence of infection.
   * Autoimmune complications including anemia or thrombocytopenia poorly responsive to corticosteroids.
   * Symptomatic or functional extranodal involvement (e.g., skin, kidney, lung, spine).
7. GCLLSG prognostic index with intermediate (3-5), high (6-10) or very high (11-14) risk scores.
8. Must have an Eastern Cooperative Oncology Group (ECOG) performance status score of ≤1.
9. All sexually active subjects with the capacity to reproduce (male and female) must use high-efficacy contraceptive methods during the course of the study. These restrictions apply for 3 months after the last dose of acalabrutinib. High-efficacy contraceptive methods include:

   * Total abstinence when consistent with the subject's typical and preferred lifestyle (periodic abstinence [e.g. calendar methods, ovulation, symptothermal and post-ovulation methods] and the withdrawal method are not acceptable contraceptive methods).
   * Female sterilisation defined as surgical hysterectomy, bilateral oophorectomy, or tubal ligation at least six weeks prior to the study treatment (a simple oophorectomy does not meet the definition of female sterilisation).
   * Male sterilisation (at least six months before screening). A man who has undergone a vasectomy must be the only partner who is a study subject.
   * Combination of two of the following methods (a+b or a+c or b+c):

     1. Use of oral, injected or implanted hormonal contraceptives, or other hormonal contraceptive methods that have a comparable efficacy (failure rate < 1%), for example, hormonal vaginal ring or transdermal hormonal contraceptive. If an oral contraceptive is used, women must use the same pill for a minimum of three months before taking the study treatment.
     2. Placement of an intrauterine device (IUD) or an intrauterine system (IUS).
     3. Barrier contraceptive methods: condom or cervical cap (cervical/vault diaphragm or cap) with foam/gel/film/spermicidal cream/vaginal suppository.
10. Female subjects of childbearing potential must have a negative serum pregnancy test at screening. Females of child bearing potential are defined as sexually mature women without prior hysterectomy or who have had any evidence of menses in the past 12 months. However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to other causes, including prior chemotherapy, anti-estrogens, or ovarian suppression.

Exclusion Criteria:

1. Prior treatment for CLL.
2. Meets any criteria for the initiation of treatment defined by the IWCLL guidelines for diagnosis and treatment of CLL (Hallek, 2018).
3. Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) and/or Hepatitis C Virus (HCV) infection and/or known history of progressive multifocal leukoencephalopathy (PML). Subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded.
4. Estimated Glomerular Filtration Rate (Cockcroft-Gault Appendix C) ≤ 40 mL/min/1.73m2.
5. Absolute neutrophil count (ANC) < 1.0 X 109/L.
6. Platelet count < 100 X 109/L.
7. Serum aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or alanine transaminase (ALT)/serum glutamate pyruvate transaminase (SGPT) >2.5 x upper limit of normal (ULN).
8. Serum total bilirubin >1.5 x ULN, except in cases of Gilbert's syndrome.
9. Prothrombin time/INR or aPTT (in the absence of Lupus anticoagulant) >2 x ULN.
10. Active bleeding, history of bleeding diathesis (e.g., hemophilia or von Willebrand disease).
11. Requires treatment with proton pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrolment to this study.
12. Unable to swallow capsules, or has disease significantly affecting gastrointestinal function that would limit absorption of oral medication.
13. Currently active, clinically significant cardiovascular disease or a history of myocardial infarction within 3 months prior to enrolment. Exception: Subjects with controlled, asymptomatic atrial fibrillation during screening can enrol on study.
14. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon) within 7 days of first dose of study drug.
15. Systemic infection that has not resolved prior to initiating study treatment in spite of adequate anti-infective therapy.
16. Pregnant or lactating females.
17. Participation in any clinical study or having taken any investigational therapy within 28 days prior to initiating study therapy.
18. Prior history of malignancies, other than CLL, unless the patient has been free of the disease for ≥ 3 years. Exceptions include the following:

    * Basal cell carcinoma of the skin
    * Squamous cell carcinoma of the skin
    * Carcinoma in situ of the cervix
    * Carcinoma in situ of the breast
    * Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b)
19. Presence of autoimmune haemolytic anaemia or autoimmune thrombocytopenia, or a positive direct antiglobulin test result.
20. Chronic use of steroids in excess of prednisone 20mg/day or its equivalent.
21. Major surgery within the last 28 days prior to registration.
22. History of stroke or intracranial hemorrhage within 6 months prior to enrolment.
23. Requires treatment with strong CYP3A4/5 Inhibitors.
24. Known history of drug-specific hypersensitivity or anaphylaxis to study drug (including active product or excipient components).
25. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of acalabrutinib, or put the study outcomes at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) | From randomization to 60 months
  EFS is defined as the time between the date of randomization and time point of symptomatic disease progression with treatment indication according to the iwCLL-Guidelines, initiation of subsequent treatment for CLL or death by any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From randomization to 60 months
  Time between the date of randomization and progression of disease or death from any cause, whichever occurs first.
Overall Survival (OS) | From randomization to 60 months
  Time between the date of randomization and death from may cause.
Time To Next Treatment (TTNT) | From randomization to 60 months
  Time from randomization until the date of initiation of subsequent treatment for CLL or death from any cause.
Objetive Response Rate (ORR) | From randomization to 60 months
  Is defined as the proportion of patients who achieve a CR (Complete Remission), CRi (CR with incomplete bone marrow recovery), nPR (nodular Partial Remission) or PR (Partial Response) over the course of the study. Patients who achieve a PR with lymphocytosis will be included in the ORR. The rate of MRD-negative disease (MRD: Minimal Residual Disease) will also be calculated. The IWCLL guidelines (Hallek, 2018) will be used to measure response in CLL.

CONTACTS AND LOCATIONS:
Overall Officials: Pau Abrisqueta Costa, MD, Principal Investigator — University Hospital of Vall d'Hebron; Francesc Bosch Albareda, MD, Principal Investigator — University Hospital of Vall d'Hebron; Carmen López Carrero, Study Chair — Fundación Pethema
Locations (8):
- Spain (8):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - ICO L´Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital Costa del Sol, Marbella
  - Hospital Universitario Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Virgen de la Salud (Complejo Hospitalario de Toledo), Toledo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrisqueta P, Pereira A, Rozman C, Aymerich M, Gine E, Moreno C, Muntanola A, Rozman M, Villamor N, Hodgson K, Campo E, Bosch F, Montserrat E. Improving survival in patients with chronic lymphocytic leukemia (1980-2008): the Hospital Clinic of Barcelona experience. Blood. 2009 Sep 3;114(10):2044-50. doi: 10.1182/blood-2009-04-214346. Epub 2009 Jun 24. PMID 19553638
- [Background] Advani RH, Buggy JJ, Sharman JP, Smith SM, Boyd TE, Grant B, Kolibaba KS, Furman RR, Rodriguez S, Chang BY, Sukbuntherng J, Izumi R, Hamdy A, Hedrick E, Fowler NH. Bruton tyrosine kinase inhibitor ibrutinib (PCI-32765) has significant activity in patients with relapsed/refractory B-cell malignancies. J Clin Oncol. 2013 Jan 1;31(1):88-94. doi: 10.1200/JCO.2012.42.7906. Epub 2012 Oct 8. PMID 23045577
- [Background] Barrientos JC, Barr PM, Flinn I, Burger JA, Salman Z, Clow F et al. Ibrutinib in combination with bendamustine and rituximab is active and tolerable in patients with relapsed/refractory CLL/SLL: final results of a phase 1b study. Blood 2013; 122: 525.[Abstract].
- [Background] Beum PV, Lindorfer MA, Beurskens F, Stukenberg PT, Lokhorst HM, Pawluczkowycz AW, Parren PW, van de Winkel JG, Taylor RP. Complement activation on B lymphocytes opsonized with rituximab or ofatumumab produces substantial changes in membrane structure preceding cell lysis. J Immunol. 2008 Jul 1;181(1):822-32. doi: 10.4049/jimmunol.181.1.822. PMID 18566448
- [Background] Bishop GA, Haxhinasto SA, Stunz LL, Hostager BS. Antigen-specific B-lymphocyte activation. Crit Rev Immunol. 2003;23(3):149-97. doi: 10.1615/critrevimmunol.v23.i3.10. PMID 14584878
- [Background] Bleeker WK, Munk ME, Mackus WJ, van den Brakel JH, Pluyter M, Glennie MJ, van de Winkel JG, Parren PW. Estimation of dose requirements for sustained in vivo activity of a therapeutic human anti-CD20 antibody. Br J Haematol. 2008 Feb;140(3):303-12. doi: 10.1111/j.1365-2141.2007.06916.x. Epub 2007 Nov 27. PMID 18045353
- [Background] Bojarczuk K, Siernicka M, Dwojak M, Bobrowicz M, Pyrzynska B, Gaj P, Karp M, Giannopoulos K, Efremov DG, Fauriat C, Golab J, Winiarska M. B-cell receptor pathway inhibitors affect CD20 levels and impair antitumor activity of anti-CD20 monoclonal antibodies. Leukemia. 2014 May;28(5):1163-7. doi: 10.1038/leu.2014.12. Epub 2014 Jan 10. No abstract available. PMID 24492323
- [Background] Bosch F, Abrisqueta P, Villamor N, Terol MJ, Gonzalez-Barca E, Ferra C, Gonzalez Diaz M, Abella E, Delgado J, Carbonell F, Garcia Marco JA, Escoda L, Ferrer S, Monzo E, Gonzalez Y, Estany C, Jarque I, Salamero O, Muntanola A, Montserrat E. Rituximab, fludarabine, cyclophosphamide, and mitoxantrone: a new, highly active chemoimmunotherapy regimen for chronic lymphocytic leukemia. J Clin Oncol. 2009 Sep 20;27(27):4578-84. doi: 10.1200/JCO.2009.22.0442. Epub 2009 Aug 24. PMID 19704063
- [Background] Brenner H, Gondos A, Pulte D. Trends in long-term survival of patients with chronic lymphocytic leukemia from the 1980s to the early 21st century. Blood. 2008 May 15;111(10):4916-21. doi: 10.1182/blood-2007-12-129379. Epub 2008 Feb 28. PMID 18309034
- [Background] Burger JA. Nurture versus nature: the microenvironment in chronic lymphocytic leukemia. Hematology Am Soc Hematol Educ Program. 2011;2011:96-103. doi: 10.1182/asheducation-2011.1.96. PMID 22160019
- [Background] Burger JA, Keating MJ, Wierda WG, Hartmann E, Hoellenriegel J, Rosin NY, de Weerdt I, Jeyakumar G, Ferrajoli A, Cardenas-Turanzas M, Lerner S, Jorgensen JL, Nogueras-Gonzalez GM, Zacharian G, Huang X, Kantarjian H, Garg N, Rosenwald A, O'Brien S. Safety and activity of ibrutinib plus rituximab for patients with high-risk chronic lymphocytic leukaemia: a single-arm, phase 2 study. Lancet Oncol. 2014 Sep;15(10):1090-9. doi: 10.1016/S1470-2045(14)70335-3. Epub 2014 Aug 20. PMID 25150798
- [Background] Burger JA, Tedeschi A, Barr PM, Robak T, Owen C, Ghia P, Bairey O, Hillmen P, Bartlett NL, Li J, Simpson D, Grosicki S, Devereux S, McCarthy H, Coutre S, Quach H, Gaidano G, Maslyak Z, Stevens DA, Janssens A, Offner F, Mayer J, O'Dwyer M, Hellmann A, Schuh A, Siddiqi T, Polliack A, Tam CS, Suri D, Cheng M, Clow F, Styles L, James DF, Kipps TJ; RESONATE-2 Investigators. Ibrutinib as Initial Therapy for Patients with Chronic Lymphocytic Leukemia. N Engl J Med. 2015 Dec 17;373(25):2425-37. doi: 10.1056/NEJMoa1509388. Epub 2015 Dec 6. PMID 26639149
- [Background] Byrd JC, Furman RR, Coutre SE, Flinn IW, Burger JA, Blum KA, Grant B, Sharman JP, Coleman M, Wierda WG, Jones JA, Zhao W, Heerema NA, Johnson AJ, Sukbuntherng J, Chang BY, Clow F, Hedrick E, Buggy JJ, James DF, O'Brien S. Targeting BTK with ibrutinib in relapsed chronic lymphocytic leukemia. N Engl J Med. 2013 Jul 4;369(1):32-42. doi: 10.1056/NEJMoa1215637. Epub 2013 Jun 19. PMID 23782158
- [Background] Byrd JC, Brown JR, O'Brien S, Barrientos JC, Kay NE, Reddy NM, Coutre S, Tam CS, Mulligan SP, Jaeger U, Devereux S, Barr PM, Furman RR, Kipps TJ, Cymbalista F, Pocock C, Thornton P, Caligaris-Cappio F, Robak T, Delgado J, Schuster SJ, Montillo M, Schuh A, de Vos S, Gill D, Bloor A, Dearden C, Moreno C, Jones JJ, Chu AD, Fardis M, McGreivy J, Clow F, James DF, Hillmen P; RESONATE Investigators. Ibrutinib versus ofatumumab in previously treated chronic lymphoid leukemia. N Engl J Med. 2014 Jul 17;371(3):213-23. doi: 10.1056/NEJMoa1400376. Epub 2014 May 31. PMID 24881631
- [Background] Byrd JC, Harrington B, O'Brien S, Jones JA, Schuh A, Devereux S, Chaves J, Wierda WG, Awan FT, Brown JR, Hillmen P, Stephens DM, Ghia P, Barrientos JC, Pagel JM, Woyach J, Johnson D, Huang J, Wang X, Kaptein A, Lannutti BJ, Covey T, Fardis M, McGreivy J, Hamdy A, Rothbaum W, Izumi R, Diacovo TG, Johnson AJ, Furman RR. Acalabrutinib (ACP-196) in Relapsed Chronic Lymphocytic Leukemia. N Engl J Med. 2016 Jan 28;374(4):323-32. doi: 10.1056/NEJMoa1509981. Epub 2015 Dec 7. PMID 26641137
- [Background] Campo E, Swerdlow SH, Harris NL, Pileri S, Stein H, Jaffe ES. The 2008 WHO classification of lymphoid neoplasms and beyond: evolving concepts and practical applications. Blood. 2011 May 12;117(19):5019-32. doi: 10.1182/blood-2011-01-293050. Epub 2011 Feb 7. PMID 21300984
- [Background] Cheson BD, Byrd JC, Rai KR, Kay NE, O'Brien SM, Flinn IW, Wiestner A, Kipps TJ. Novel targeted agents and the need to refine clinical end points in chronic lymphocytic leukemia. J Clin Oncol. 2012 Aug 10;30(23):2820-2. doi: 10.1200/JCO.2012.43.3748. Epub 2012 Jul 9. No abstract available. PMID 22778323
- [Background] Chiorazzi N, Rai KR, Ferrarini M. Chronic lymphocytic leukemia. N Engl J Med. 2005 Feb 24;352(8):804-15. doi: 10.1056/NEJMra041720. No abstract available. PMID 15728813
- [Background] Coiffier B, Lepretre S, Pedersen LM, Gadeberg O, Fredriksen H, van Oers MH, Wooldridge J, Kloczko J, Holowiecki J, Hellmann A, Walewski J, Flensburg M, Petersen J, Robak T. Safety and efficacy of ofatumumab, a fully human monoclonal anti-CD20 antibody, in patients with relapsed or refractory B-cell chronic lymphocytic leukemia: a phase 1-2 study. Blood. 2008 Feb 1;111(3):1094-100. doi: 10.1182/blood-2007-09-111781. Epub 2007 Nov 14. PMID 18003886
- [Background] Craxton A, Jiang A, Kurosaki T, Clark EA. Syk and Bruton's tyrosine kinase are required for B cell antigen receptor-mediated activation of the kinase Akt. J Biol Chem. 1999 Oct 22;274(43):30644-50. doi: 10.1074/jbc.274.43.30644. PMID 10521450
- [Background] Da Roit F, Engelberts PJ, Taylor RP, Breij EC, Gritti G, Rambaldi A, Introna M, Parren PW, Beurskens FJ, Golay J. Ibrutinib interferes with the cell-mediated anti-tumor activities of therapeutic CD20 antibodies: implications for combination therapy. Haematologica. 2015 Jan;100(1):77-86. doi: 10.3324/haematol.2014.107011. Epub 2014 Oct 24. PMID 25344523
- [Background] Dighiero G, Maloum K, Desablens B, Cazin B, Navarro M, Leblay R, Leporrier M, Jaubert J, Lepeu G, Dreyfus B, Binet JL, Travade P. Chlorambucil in indolent chronic lymphocytic leukemia. French Cooperative Group on Chronic Lymphocytic Leukemia. N Engl J Med. 1998 May 21;338(21):1506-14. doi: 10.1056/NEJM199805213382104. PMID 9593789
- [Background] Eichhorst BF, Busch R, Hopfinger G, Pasold R, Hensel M, Steinbrecher C, Siehl S, Jager U, Bergmann M, Stilgenbauer S, Schweighofer C, Wendtner CM, Dohner H, Brittinger G, Emmerich B, Hallek M; German CLL Study Group. Fludarabine plus cyclophosphamide versus fludarabine alone in first-line therapy of younger patients with chronic lymphocytic leukemia. Blood. 2006 Feb 1;107(3):885-91. doi: 10.1182/blood-2005-06-2395. Epub 2005 Oct 11. PMID 16219797
- [Background] Flinn IW, Neuberg DS, Grever MR, Dewald GW, Bennett JM, Paietta EM, Hussein MA, Appelbaum FR, Larson RA, Moore DF Jr, Tallman MS. Phase III trial of fludarabine plus cyclophosphamide compared with fludarabine for patients with previously untreated chronic lymphocytic leukemia: US Intergroup Trial E2997. J Clin Oncol. 2007 Mar 1;25(7):793-8. doi: 10.1200/JCO.2006.08.0762. Epub 2007 Feb 5. PMID 17283364
- [Background] Flinn IW, Byrd JC, Morrison C, Jamison J, Diehl LF, Murphy T, Piantadosi S, Seifter E, Ambinder RF, Vogelsang G, Grever MR. Fludarabine and cyclophosphamide with filgrastim support in patients with previously untreated indolent lymphoid malignancies. Blood. 2000 Jul 1;96(1):71-5. PMID 10891432
- [Background] Gribben JG, O'Brien S. Update on therapy of chronic lymphocytic leukemia. J Clin Oncol. 2011 Feb 10;29(5):544-50. doi: 10.1200/JCO.2010.32.3865. Epub 2011 Jan 10. PMID 21220603
- [Background] Gururajan M, Jennings CD, Bondada S. Cutting edge: constitutive B cell receptor signaling is critical for basal growth of B lymphoma. J Immunol. 2006 May 15;176(10):5715-9. doi: 10.4049/jimmunol.176.10.5715. PMID 16670274
- [Background] Hagenbeek A, Gadeberg O, Johnson P, Pedersen LM, Walewski J, Hellmann A, Link BK, Robak T, Wojtukiewicz M, Pfreundschuh M, Kneba M, Engert A, Sonneveld P, Flensburg M, Petersen J, Losic N, Radford J. First clinical use of ofatumumab, a novel fully human anti-CD20 monoclonal antibody in relapsed or refractory follicular lymphoma: results of a phase 1/2 trial. Blood. 2008 Jun 15;111(12):5486-95. doi: 10.1182/blood-2007-10-117671. Epub 2008 Apr 4. PMID 18390837
- [Background] Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, Hillmen P, Keating M, Montserrat E, Chiorazzi N, Stilgenbauer S, Rai KR, Byrd JC, Eichhorst B, O'Brien S, Robak T, Seymour JF, Kipps TJ. iwCLL guidelines for diagnosis, indications for treatment, response assessment, and supportive management of CLL. Blood. 2018 Jun 21;131(25):2745-2760. doi: 10.1182/blood-2017-09-806398. Epub 2018 Mar 14. PMID 29540348
- [Background] Hallek M, Fischer K, Fingerle-Rowson G, Fink AM, Busch R, Mayer J, Hensel M, Hopfinger G, Hess G, von Grunhagen U, Bergmann M, Catalano J, Zinzani PL, Caligaris-Cappio F, Seymour JF, Berrebi A, Jager U, Cazin B, Trneny M, Westermann A, Wendtner CM, Eichhorst BF, Staib P, Buhler A, Winkler D, Zenz T, Bottcher S, Ritgen M, Mendila M, Kneba M, Dohner H, Stilgenbauer S; International Group of Investigators; German Chronic Lymphocytic Leukaemia Study Group. Addition of rituximab to fludarabine and cyclophosphamide in patients with chronic lymphocytic leukaemia: a randomised, open-label, phase 3 trial. Lancet. 2010 Oct 2;376(9747):1164-74. doi: 10.1016/S0140-6736(10)61381-5. PMID 20888994
- [Background] Herman SE, Gordon AL, Hertlein E, Ramanunni A, Zhang X, Jaglowski S, Flynn J, Jones J, Blum KA, Buggy JJ, Hamdy A, Johnson AJ, Byrd JC. Bruton tyrosine kinase represents a promising therapeutic target for treatment of chronic lymphocytic leukemia and is effectively targeted by PCI-32765. Blood. 2011 Jun 9;117(23):6287-96. doi: 10.1182/blood-2011-01-328484. Epub 2011 Mar 21. PMID 21422473
- [Background] Hoechstetter MA, Busch R, Eichhorst B, Buhler A, Winkler D, Eckart MJ, Vehling-Kaiser U, Schimke H, Jager U, Hurtz HJ, Hopfinger G, Hartmann F, Fuss H, Abenhardt W, Blau I, Freier W, Muller L, Goebeler M, Wendtner CM, Bahlo J, Fischer K, Bentz M, Emmerich B, Dohner H, Hallek M, Stilgenbauer S. Early, risk-adapted treatment with fludarabine in Binet stage A chronic lymphocytic leukemia patients: results of the CLL1 trial of the German CLL study group. Leukemia. 2017 Dec;31(12):2833-2837. doi: 10.1038/leu.2017.246. Epub 2017 Aug 14. No abstract available. PMID 28804126
- [Background] Honigberg LA, Smith AM, Sirisawad M, Verner E, Loury D, Chang B, Li S, Pan Z, Thamm DH, Miller RA, Buggy JJ. The Bruton tyrosine kinase inhibitor PCI-32765 blocks B-cell activation and is efficacious in models of autoimmune disease and B-cell malignancy. Proc Natl Acad Sci U S A. 2010 Jul 20;107(29):13075-80. doi: 10.1073/pnas.1004594107. Epub 2010 Jul 6. PMID 20615965
- [Background] Kohrt HE, Sagiv-Barfi I, Rafiq S, Herman SE, Butchar JP, Cheney C, Zhang X, Buggy JJ, Muthusamy N, Levy R, Johnson AJ, Byrd JC. Ibrutinib antagonizes rituximab-dependent NK cell-mediated cytotoxicity. Blood. 2014 Mar 20;123(12):1957-60. doi: 10.1182/blood-2014-01-547869. No abstract available. PMID 24652965
- [Background] Kuppers R. Mechanisms of B-cell lymphoma pathogenesis. Nat Rev Cancer. 2005 Apr;5(4):251-62. doi: 10.1038/nrc1589. PMID 15803153
- [Background] Langerbeins P, Bahlo J, Rhein C, Cramer P, Pflug N, Fischer K, Stilgenbauer S, Kreuzer KA, Wendtner CM, Eichhorst B, Hallek M. The CLL12 trial protocol: a placebo-controlled double-blind Phase III study of ibrutinib in the treatment of early-stage chronic lymphocytic leukemia patients with risk of early disease progression. Future Oncol. 2015;11(13):1895-903. doi: 10.2217/fon.15.95. PMID 26161926
- [Background] Meeker T, Lowder J, Cleary ML, Stewart S, Warnke R, Sklar J, Levy R. Emergence of idiotype variants during treatment of B-cell lymphoma with anti-idiotype antibodies. N Engl J Med. 1985 Jun 27;312(26):1658-65. doi: 10.1056/NEJM198506273122602. PMID 3923352
- [Background] Miller MD, Paradis CF, Houck PR, Mazumdar S, Stack JA, Rifai AH, Mulsant B, Reynolds CF 3rd. Rating chronic medical illness burden in geropsychiatric practice and research: application of the Cumulative Illness Rating Scale. Psychiatry Res. 1992 Mar;41(3):237-48. doi: 10.1016/0165-1781(92)90005-n. PMID 1594710
- [Background] National Comprehensive Cancer Network (NCCN). NCCN Clinical Practice Guidelines in Oncology (NCCN Guidelines) Non-Hodgkin's Lymphomas. Version I.2012. NCCN.org
- [Background] O'Brien SM, Kantarjian HM, Cortes J, Beran M, Koller CA, Giles FJ, Lerner S, Keating M. Results of the fludarabine and cyclophosphamide combination regimen in chronic lymphocytic leukemia. J Clin Oncol. 2001 Mar 1;19(5):1414-20. doi: 10.1200/JCO.2001.19.5.1414. PMID 11230486
- [Background] O'Brien S, Furman RR, Coutre SE, Sharman JP, Burger JA, Blum KA, Grant B, Richards DA, Coleman M, Wierda WG, Jones JA, Zhao W, Heerema NA, Johnson AJ, Izumi R, Hamdy A, Chang BY, Graef T, Clow F, Buggy JJ, James DF, Byrd JC. Ibrutinib as initial therapy for elderly patients with chronic lymphocytic leukaemia or small lymphocytic lymphoma: an open-label, multicentre, phase 1b/2 trial. Lancet Oncol. 2014 Jan;15(1):48-58. doi: 10.1016/S1470-2045(13)70513-8. Epub 2013 Dec 10. PMID 24332241
- [Background] Pawluczkowycz AW, Beurskens FJ, Beum PV, Lindorfer MA, van de Winkel JG, Parren PW, Taylor RP. Binding of submaximal C1q promotes complement-dependent cytotoxicity (CDC) of B cells opsonized with anti-CD20 mAbs ofatumumab (OFA) or rituximab (RTX): considerably higher levels of CDC are induced by OFA than by RTX. J Immunol. 2009 Jul 1;183(1):749-58. doi: 10.4049/jimmunol.0900632. Epub 2009 Jun 17. PMID 19535640
- [Background] Petro JB, Rahman SM, Ballard DW, Khan WN. Bruton's tyrosine kinase is required for activation of IkappaB kinase and nuclear factor kappaB in response to B cell receptor engagement. J Exp Med. 2000 May 15;191(10):1745-54. doi: 10.1084/jem.191.10.1745. PMID 10811867
- [Background] Petro JB, Khan WN. Phospholipase C-gamma 2 couples Bruton's tyrosine kinase to the NF-kappaB signaling pathway in B lymphocytes. J Biol Chem. 2001 Jan 19;276(3):1715-9. doi: 10.1074/jbc.M009137200. Epub 2000 Oct 19. PMID 11042193
- [Background] Pflug N, Bahlo J, Shanafelt TD, Eichhorst BF, Bergmann MA, Elter T, Bauer K, Malchau G, Rabe KG, Stilgenbauer S, Dohner H, Jager U, Eckart MJ, Hopfinger G, Busch R, Fink AM, Wendtner CM, Fischer K, Kay NE, Hallek M. Development of a comprehensive prognostic index for patients with chronic lymphocytic leukemia. Blood. 2014 Jul 3;124(1):49-62. doi: 10.1182/blood-2014-02-556399. Epub 2014 May 5. PMID 24797299
- [Background] Ponader S, Chen SS, Buggy JJ, Balakrishnan K, Gandhi V, Wierda WG, Keating MJ, O'Brien S, Chiorazzi N, Burger JA. The Bruton tyrosine kinase inhibitor PCI-32765 thwarts chronic lymphocytic leukemia cell survival and tissue homing in vitro and in vivo. Blood. 2012 Feb 2;119(5):1182-9. doi: 10.1182/blood-2011-10-386417. Epub 2011 Dec 16. PMID 22180443
- [Background] Satterthwaite AB, Witte ON. The role of Bruton's tyrosine kinase in B-cell development and function: a genetic perspective. Immunol Rev. 2000 Jun;175:120-7. PMID 10933597
- [Background] Shaffer AL, Rosenwald A, Staudt LM. Lymphoid malignancies: the dark side of B-cell differentiation. Nat Rev Immunol. 2002 Dec;2(12):920-32. doi: 10.1038/nri953. PMID 12461565
- [Background] Smith TJ, Khatcheressian J, Lyman GH, Ozer H, Armitage JO, Balducci L, Bennett CL, Cantor SB, Crawford J, Cross SJ, Demetri G, Desch CE, Pizzo PA, Schiffer CA, Schwartzberg L, Somerfield MR, Somlo G, Wade JC, Wade JL, Winn RJ, Wozniak AJ, Wolff AC. 2006 update of recommendations for the use of white blood cell growth factors: an evidence-based clinical practice guideline. J Clin Oncol. 2006 Jul 1;24(19):3187-205. doi: 10.1200/JCO.2006.06.4451. Epub 2006 May 8. PMID 16682719
- [Background] Spaargaren M, Beuling EA, Rurup ML, Meijer HP, Klok MD, Middendorp S, Hendriks RW, Pals ST. The B cell antigen receptor controls integrin activity through Btk and PLCgamma2. J Exp Med. 2003 Nov 17;198(10):1539-50. doi: 10.1084/jem.20011866. Epub 2003 Nov 10. PMID 14610042
- [Background] Surveillance Epidemiology and End Results (SEER), NCI, US National Institutes of Health, Fast Stats; Statistics Stratified by Cancer Site, 2010.
- [Background] Tam CS, O'Brien S, Wierda W, Kantarjian H, Wen S, Do KA, Thomas DA, Cortes J, Lerner S, Keating MJ. Long-term results of the fludarabine, cyclophosphamide, and rituximab regimen as initial therapy of chronic lymphocytic leukemia. Blood. 2008 Aug 15;112(4):975-80. doi: 10.1182/blood-2008-02-140582. Epub 2008 Apr 14. PMID 18411418
- [Background] Teeling JL, French RR, Cragg MS, van den Brakel J, Pluyter M, Huang H, Chan C, Parren PW, Hack CE, Dechant M, Valerius T, van de Winkel JG, Glennie MJ. Characterization of new human CD20 monoclonal antibodies with potent cytolytic activity against non-Hodgkin lymphomas. Blood. 2004 Sep 15;104(6):1793-800. doi: 10.1182/blood-2004-01-0039. Epub 2004 Jun 1. PMID 15172969
- [Background] Teeling JL, Mackus WJ, Wiegman LJ, van den Brakel JH, Beers SA, French RR, van Meerten T, Ebeling S, Vink T, Slootstra JW, Parren PW, Glennie MJ, van de Winkel JG. The biological activity of human CD20 monoclonal antibodies is linked to unique epitopes on CD20. J Immunol. 2006 Jul 1;177(1):362-71. doi: 10.4049/jimmunol.177.1.362. PMID 16785532
- [Background] Tomlinson MG, Woods DB, McMahon M, Wahl MI, Witte ON, Kurosaki T, Bolen JB, Johnston JA. A conditional form of Bruton's tyrosine kinase is sufficient to activate multiple downstream signaling pathways via PLC Gamma 2 in B cells. BMC Immunol. 2001;2:4. doi: 10.1186/1471-2172-2-4. Epub 2001 Jun 8. PMID 11410123
- [Background] Welch HG, Albertsen PC, Nease RF, Bubolz TA, Wasson JH. Estimating treatment benefits for the elderly: the effect of competing risks. Ann Intern Med. 1996 Mar 15;124(6):577-84. doi: 10.7326/0003-4819-124-6-199603150-00007. PMID 8597322
- [Background] Wierda WG, Kipps TJ, Mayer J, Stilgenbauer S, Williams CD, Hellmann A, Robak T, Furman RR, Hillmen P, Trneny M, Dyer MJ, Padmanabhan S, Piotrowska M, Kozak T, Chan G, Davis R, Losic N, Wilms J, Russell CA, Osterborg A; Hx-CD20-406 Study Investigators. Ofatumumab as single-agent CD20 immunotherapy in fludarabine-refractory chronic lymphocytic leukemia. J Clin Oncol. 2010 Apr 1;28(10):1749-55. doi: 10.1200/JCO.2009.25.3187. Epub 2010 Mar 1. PMID 20194866
- [Background] Wierda WG, Kipps TJ, Durig J, Griskevicius L, Stilgenbauer S, Mayer J, Smolej L, Hess G, Griniute R, Hernandez-Ilizaliturri FJ, Padmanabhan S, Gorczyca M, Chang CN, Chan G, Gupta I, Nielsen TG, Russell CA; 407 Study Investigators. Chemoimmunotherapy with O-FC in previously untreated patients with chronic lymphocytic leukemia. Blood. 2011 Jun 16;117(24):6450-8. doi: 10.1182/blood-2010-12-323980. Epub 2011 Apr 15. PMID 21498674